CLINICAL TRIAL: NCT01273350
Title: Physician I.D.E. G#040160; Low Risk Carotid Stenting Study Using Bivalirudin at PinnacleHealth Hospitals and Holy Spirit Hospital
Brief Title: A Prospective, Non-Randomized, Evaluation of Low-Risk Patients Undergoing Carotid Stenting With ANgiomax (Bivalirudin)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SPSI d.b.a Capital Cardiovascular Associates (Other)
Responsible Party: Principal Investigator, Rajesh Dave, MD, Chief Medical Executive Holy Spirit Cardiovascular Institute, SPSI d.b.a Capital Cardiovascular Associates
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Physician IDE G # 040160
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Carotid Stenosis
Keywords: internal carotid artery; common carotid artery; bruit; tia
MeSH Terms: conditions — Carotid Stenosis; Ischemic Attack, Transient | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Other): Single arm observational study looking at a "low risk" cohort of individuals with carotid stenosis
  Interventions: Device: Carotid PTA and stenting

INTERVENTIONS:
Device: Carotid PTA and stenting — Percutaneous interventional treatment of carotid artery stenosis using XACT carotid artery stent and emboshield protection system with bivalirudin as the procedural anticoagulant

SUMMARY:
Prospective, non-randomized, single-center cohort study treating internal carotid artery stenosis using the Xact Carotid Artery Stent and emboshield distal protection system in conjunction with bivalirudin as the procedural anticoagulation

DETAILED DESCRIPTION:
Primary objective is to evaluate the safety and feasibility of the XACT stent and emboshield with Angiomax as the procedural anticoagulant.

Primary safety endpoint is the occurrence of Major Adverse Events, defined as death, myocardial infarction (Q or non Q wave), and from target revascularization at one year

ELIGIBILITY:
Inclusion Criteria:

* Patient (male or non-pregnant female)must be > than or= 18
* Qualifying non-invasive test (ultrasound or MRA) was performed less than 60 days prior to study entry. Carotid duplex study revealed:

  * Stenosis > or = to 50% in symptomatic patients
  * Stenosis > or = to 60% in asymptomatic patients
* Target lesion may be in the common or internal carotid artery and is amenable to treatment with angioplasty and stenting
* Patients taking warfarin may be included if their dosage is reduced before the procedure to result in an INR of 1.5 or less and a Prothrombin time of 15 seconds. Warfarin may be started after the procedure.
* Female patients of childbearing potential must have a documented negative pregnancy test during index hospitalization
* Patient or legally authorized representative must sign a written informed consent, prior to the procedure, using a form that is approved by the local institutional review board or medical ethics committee

Exclusion Criteria: (Patients will be excluded from the study if ANY of the following conditions are present)

* There is total occlusion of the target carotid artery treatment site.
* The patient has an allergy or contraindication to aspirin, ticlopidine, clopidogrel, bivalirudin, nickel, titanium, or a sensitivity to contrast media, which cannot adequately pre-medicated.
* The subject has a platlet count< 100,000 cells/mm3 or 700,000 cells/mm3 or a WBC of < 3,000 cells/mm3.
* Stroke within 7 days prior to the procedure
* NIH stroke score > or = to 15 within 7 days prior to the procedure
* The patient has experienced a significant GI bleed within 6 months prior to study procedure
* The patient has active internal bleeding
* The patient has had major surgery or serious trauma within 6 weeks before enrollment
* The patient has excessive peripheral vascular disease that precludes safe sheath insertion
* The patient has had an intracranial hemorrhage, hemorrhagic stroke, major stroke or any stroke within one week of index procedure
* The patient has concurrent emboligenic cardiovascular disease not adequately treated with anticoagulant therapy
* The patient is on renal dialysis
* The patient has had low molecular weight heparin (LMWH) administered within 8 hours or less, prior to the procedure
* Severe hypertension not adequately controlled by antihypertensive therapy at the time of study entry(BP> 180/110mmHG)
* The patient is unable or unwilling to cooperate with the study follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2004-10; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Major adverse events, defined as death, ipsilateral stroke, myocardial infarction,(Q and non-Q wave) or major bleeding as 30 days post procedure | 30 days

SECONDARY OUTCOMES:
Freedom from vascular complications ;Acute success defined by lesion, device, and procedural success; Freedom from any death, stroke MI (Q, non-Q wave), and from target lesion revascularization at one year | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh M Dave, MD, Principal Investigator — Spirit Physician Services Inc. d.b.a.Capital Cardiovascular Associates @ PinnacleHealth Hospitals; Holy Spirit Hospital
Locations (1):
- Spirit Physycian Services Inc.d.b.a Capital Cardiovascular Associates, Camp Hill, Pennsylvania, United States